CLINICAL TRIAL: NCT04374240
Title: Phase I Trial of Replicative Defective Type 5 Adenovirus Vector Expressing Nitroreductase & GMCSF Given Via Trans-perineal Template-guided Intra-prostatic Injection Followed by iv CB1954 in Locally Relapsed Prostate Cancer Patients
Brief Title: A Clinical Trial of AdNRGM Plus CB1954 in Prostate Cancer
Acronym: AdUP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Janssen, LP (Industry); Department of Health, United Kingdom (Other Government); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_06-226; ISRCTN06254734 (Registry Identifier: ISRCTN); 2007-007041-13 (EudraCT Number)
Record Dates: First submitted 2016-03-01; First posted 2020-05-05 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer
Keywords: adenovirus
MeSH Terms: conditions — Prostatic Neoplasms; Adenoviridae Infections | interventions — tretazicar

STUDY DESIGN:
Intervention Model Description: AdNRGM plus CB1954
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdNRGM followed on day 2 by CB1954 (Experimental): The proposed dose levels for AdNRGM are 10^10, 3x10^10, 10^11, 3x10^11, 10^12 vp while the prodrug CB1954 will be given at a standard dose of 24 mg/m^2
  Interventions: Genetic: AdNRGM

INTERVENTIONS:
Genetic: AdNRGM — AdNRGM is an E1-E3 deleted, replication deficient type 5 adenovirus which contains the E. coli NTR gene regulated by the CMV promoter, an internal ribosomal entry site (IRES) and the human GMCSF gene.
  CB1954 [5-(aziridin-1-yl)-2,4-dinitrobenzamide]
  Other Names: CB1954

SUMMARY:
This is an open label, non-randomised, phase I, sequential group trial which will explore the safety and tolerability of ascending doses of AdNRGM, in combination with CB1954. Five groups of 3 patients each will be treated with escalating doses of AdNRGM (10^10, 3x10^10, 10^11, 3x10^11, 10^12 vp) followed 2 days later by intravenous CB1954 at a fixed dose (24mg/m^2). To ensure the coverage of the whole prostate the vector will be delivered by multiple, template-guided trans-perineal injections using an adaptation of standard prostate brachytherapy technique. Dose escalation will be dependent on safety and tolerability; at each dose-level, if dose-limiting toxicity (DLT) is seen in one patient, the cohort will be expanded to a maximum of 6 patients. If DLT is then observed in a second patient at that dose, no further patients will be recruited and the previous (lower) dose-level will be defined as the maximum tolerated dose (MTD). If DLT is seen in 0/3 or just 1/6 patients, dose escalation may continue.

DETAILED DESCRIPTION:
Background and Rationale:

Locally relapsed prostate cancer presents an attractive target for gene therapy because the tumour remains localised to the prostate or to the surrounding tissue for a long phase of the disease. Also the delivery of gene therapy vectors to the prostate is straightforward using either ultrasound-guided, trans-rectal injection or adapting methods developed for brachytherapy, to deliver multiple, template-guided trans-perineal injections to achieve saturation coverage of the prostate. Several gene therapy and gene-immunotherapy strategies have been tested in patients with locally relapsed or metastatic prostate cancer, including Virus Directed Enzyme Prodrug Therapy (VDEPT), Conditionally Replicating Adenoviruses (CRAds) and GMCSF based immune stimulation. These treatments were well tolerated and showed some evidence of anti-tumour activity.

The nitroreductase/CB1954 VDEPT system:

The nitroreductase/CB1954 system employs E. coli nitroreductase (NTR) as the prodrug activating enzyme, and CB1954 as the prodrug to be activated. To exploit this system a an E1-E3 deleted, replication-defective human adenovirus (Ad5) designated CTL102 which contains the NTR gene under the control of the cytomegalovirus (CMV) promoter was previously generated. CTL102 was able to infect cancer cells and to induce NTR expression in vitro, in addition NTR expressing cells are sensitised to CB1954. Experiments carried out in animal models demonstrated that NTR expression could be detected in prostate cancer xenografts injected with CTL102 and that growth of the xenografts was inhibited by intratumoural injection of CTL102 followed 2 days later by intra peritoneal administration of CB1954.

CB1954 prodrug conversion and clinical development:

CB1954 [5-(aziridin-1-yl)-2,4-dinitrobenzamide] is a weak alkylating agent that is reduced by the rat nitroreductase enzyme DT diaphorase to a potent, bifunctional alkylating agent (5-(aziridin-1-yl)-4-hydroxylamino-2-nitrobenzamide) that cross-links DNA and is able to kill both dividing and non-dividing cells. The human and murine forms of DT diaphorase are deficient in this reaction. A nitroreductase enzyme encoded by the nfsB gene of E. coli was found to perform the same reduction 60 to 100-fold faster than the rat DT diaphorase, and this is the enzyme (NTR) encoded in CTL102 and AdNRGM.

A phase I pharmacokinetic trial of CB1954 defined its maximum tolerated dose (MTD), dose-limiting toxicities and plasma concentration-time profile. Ten cohorts of three patients each were treated with CB1954 at dose levels of 3mg/m2 to 37.5 mg/m^2. No marrow suppression, nephrotoxicity or alopecia was observed. Dose limiting toxicities (one grade 4 diarrhoea and two grade 2 hepatic toxicity) were seen at 37.5 mg/m^2; other toxicities included nausea, vomiting, anorexia and fatigue. Side effects recorded at 24 mg/m^2 were grade 3 nausea and fatigue, therefore this dose was recommended as the standard dose for future clinical trials. A clouding of the lens of the eye, also known as cataract, occurred in a few animals given the CB1954 drug. The Investigators believe this change is highly unlikely to occur in humans and none of the patients who were treated with this drug in previous clinical trials has suffered from this complication.

Prostate cancer trial:

A phase I/II clinical trial of CTL102/CB1954 was completed in men with prostate cancer. In the first stage of the trial 20 patients who were scheduled for radical prostatectomy received CTL102 alone, via intraprostatic injection, prior to surgery. Objectives of this part of the study were safety, tolerability and level of NTR expression. Immunohistochemistry demonstrated NTR staining of the glandular epithelium of the tumour and of the normal prostate tissue at all dose levels which were used (1x10^10 to 1x10^12 virus particles). Expression of NTR was found in 30-50% of the prostate specimen slides and appeared to increase when using higher vector doses or multiple injections, however there was no statistically significant relationship between virus dose and extent of NTR expression. Gene therapy was well tolerated, although one patient who received 5x10^10 vp had a DLT (transient bilirubin increase). The cohort was therefore expanded but no other DLT was observed and dose escalation could be resumed. (The DLT was subsequently attributed to a post-operative myocardial infarction.) Other adverse events were transient grade 3 lymphopaenia (3 patients) and grade 2 hepatic enzymes increase (4 patients). There were no treatment-related serious adverse events.

Our data show that the intraprostatic injection of CTL102 followed by intravenous CB1954 is safe and well tolerated11. CTL102 was able to induce NTR expression and the CTL102/CB1954 treatment provided early indications of activity. However, the overall anti-tumour efficacy of this approach was sub-optimal, with only two patients showing a PSA decrease >50% and viable tumour cells still present in post-treatment biopsies. It is likely that the relatively small fraction of tumour cells expressing NTR, and their localised distribution was responsible for the limited anti-tumour activity of CTL102/CB1954. In order to increase efficacy the current clinical trial has incorporated two significant improvements:

1. To achieve better distribution of the vector throughout the prostate the vector will be administered using an adaptation of the technique of prostate brachytherapy, via multiple template-guided trans-perineal injections.
2. To increase efficacy VDEPT with GMCSF based immune stimulation, using an E1,E3-deleted, replication defective adenovirus (AdNRGM) expressing both NTR and human GMCSF will be combined.

The proposed dose levels for AdNRGM are 10^10, 3x10^10, 10^11, 3x10^11, 10^12 vp while the prodrug CB1954 will be given at a standard dose of 24 mg/m^2. In vitro experiments allow us to estimate that 1 x 10^10 vp of AdNRGM is likely to result in production of 5 - 25 µg GMCSF/24 h. Clinical trials of GMCSF have used single doses of 500 µg, or repeated doses of up to 250 µg/m^2. The Investigators consider that a starting dose of 1 x 10^10 vp therefore provides a sufficient safety margin for GMCSF production. The fixed dose or 24 mg/m^2 CB1954 is the dose recommended following an initial dose-escalation trial of CB1954 alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with biopsy-proven local recurrence of prostate cancer following radical radiotherapy and a rising PSA with or without androgen suppression with antiandrogens or LHRH agonist/antagonist therapy or after bilateral orchidectomy. A rising PSA is defined as 2 increases over 3 or 4 readings over a minimum period of 6 weeks, with time-points separated by at least 2 weeks. If the patient is on antiandrogens or LHRH agonist/antagonist therapy, this therapy should be continued.
* Life expectancy greater than 3 months.
* Aged at least 18 years.
* Written informed consent.
* World Health Organisation (WHO) performance status of 0-1.
* PSA value ≥ 2 and ≤ 100 ng/ml at study entry.
* Adequate hepatic function (i.e. bilirubin, AST, ALT all < 1.5 x upper limit of normal for Institution).
* Normal renal function (<1.25 x upper normal limit for the Institution).
* Adequate haematological function (i.e. haemoglobin > 10g/dl, WCC > 3x109/l, platelets > 150x10^9/l) and normal clotting (INR and APTT <1.2).
* Patients must agree not to father a child within 12 months following AdNRGM administration, and must use at least two methods of contraception, one of which is barrier, starting from the time of AdNRGM administration for at least 12 months.
* No known immuno-incompetence.

Exclusion Criteria:

* Patients with a prostate or abnormal focus which is deemed clinically unsuitable for trans-perineal template-guided injection.
* Patients who have previously been treated with prostate brachytherapy.
* Patients who have previously been treated with AdNRGM and CB1954; or who have been administered any other human adenovirus type 5 vector within the last 5 years.
* Patients who have received chemotherapy, radiotherapy or immunotherapy within 28 days of study entry.
* Acute active infection (viral, bacterial, or fungal) which requires specific therapy.
* Chronic hepatitis B or C infection, HIV positive patients. (Patients will be tested for HBV/HCV, but not HIV).
* Concurrent severe medical illnesses incompatible with the treatment including psychiatric pathology likely to affect protocol compliance.
* Tumours of other organs or tissues of high malignant potential still active or treated radically less than 3 years before (except that successfully treated, non-metastatic skin cancers or non-muscle invasive bladder cancers are not an exclusion criterion).
* Concurrent corticosteroids, or any medication known to have significant immunosuppressive action.
* Patients unable to travel for regular hospital assessments.
* Evidence of adenovirus infection and/or shedding at baseline.
* Clinical judgement by the Investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of escalating doses of AdNRGM, followed by iv CB1954 determined by assessing local effects on tumour etc. and number of participants with treatment related adverse events by CTCAE v4.0 | 12 months
  * Safety will be assessed in terms of local effects on the tumour, the prostate gland and the lower urinary tract as well as in terms of systemic effects. The data will be summarised descriptively.
  * Adverse events and side effects will be determined as changes of the relevant clinical parameters as well as changes of haematological and clinical biochemistry data.

SECONDARY OUTCOMES:
Measuring PSA levels following treatment with AdNRGM and CB1954 | 12 months
  Changes in the level (ng/ml) of the serum PSA will be measured in to provide an indication of changes in tumour burden, growth rate and possible anti-tumour activity of the treatment.

OTHER OUTCOMES:
To assess the evidence for local tumour destruction, and immune infiltration, in tumour biopsies taken after the treatment | 8 weeks post treatment
  Treatment-induced immune responses will be assessed by measurement of T cell responses to prostate cancer antigens in blood samples collected at baseline and at intervals (2, 3, 4, and 8 weeks) following treatment.
To investigate changes in cellular immune response to prostate cancer antigens following treatment with AdNRGM and CB1954 | 12 months
  Evidence of tumour destruction and immune infiltration will be assessed by looking at patterns of tissue damage, residual tumour tissue and immune cell infiltrates detected by immunohistochemistry in post treatment prostate biopsies .

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Patel, FRCS Ed, Principal Investigator — University of Birmingham
Locations (1):
- Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel P, Young JG, Mautner V, Ashdown D, Bonney S, Pineda RG, Collins SI, Searle PF, Hull D, Peers E, Chester J, Wallace DM, Doherty A, Leung H, Young LS, James ND. A phase I/II clinical trial in localized prostate cancer of an adenovirus expressing nitroreductase with CB1954 [correction of CB1984]. Mol Ther. 2009 Jul;17(7):1292-9. doi: 10.1038/mt.2009.80. Epub 2009 Apr 14. PMID 19367257
- See also: Trial Website — https://www.birmingham.ac.uk/research/crctu/trials/adUP/index.aspx